CLINICAL TRIAL: NCT02496988
Title: A Study of CIK in Combination With Temozolomide With and Without Radiation in Adults With Advanced Malignant Gliomas
Brief Title: Effect of Cytokine-induced Killer Cells for Advanced Malignant Gliomas
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: GLICIK002
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Cytokine-Induced Killer Cells; Advanced Milignant Gliomas
Keywords: Cytokine-Induced Killer Cells; Milignant Gliomas; Temozolomide
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temozolomide (Other): Capsules supplied in 5-mg, 20-mg, 100-mg, 140-mg, 180-mg, and 250-mg strengths; dosed at 200 mg/m2/day for 5 consecutive days, repeated every 28 days
  Interventions: Drug: Temozolomide
- Temozolomide+CIK (Other): Autologous cytokine-induced killer cells were transfer via venous one week after Temozolomide treat
  Interventions: Biological: CIK

INTERVENTIONS:
Drug: Temozolomide — Capsules supplied in 5-mg, 20-mg, 100-mg, 140-mg, 180-mg, and 250-mg strengths; dosed at 200 mg/m2/day for 5 consecutive days, repeated every 28 days
  Arms: Temozolomide
Biological: CIK — The patients received autologous cytokine-induced killer cells transfusion one week after Temozolomide treat
  Arms: Temozolomide+CIK

SUMMARY:
The purpose of this study is to determine whether combining of Temozolomide and cytokine-induced killer cells (CIK) transfusion can prolong survival of patients with Advanced Malignant Gliomas. The effectiveness and safety of CIK cells for the treatment of Malignant Glioma is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented histologically confirmed primary grade 4 advanced malignant glioma.
* No more than 3 prior relapses or prior systemic treatments.
* Recurrent disease documented by MRI after prior therapy.
* Must have at least one site of bidimensionally measurable disease:

archived tissue from the initial diagnosis of advanced malignant glioma or upon transformation to advanced malignant glioma are available for central review within approximately 4 weeks after enrollment.

* Completed at least one full cycle of temozolomide of 200 mg/m2/day administered on Days 1-5 of a 28-day cycle, without unacceptable toxicity or progression.
* Karnofsky performance status of 60 or more. Adequate organ and bone marrow function as defined by hematological and serum chemistry limits.
* At least 18 years old.
* Both men and women must practice adequate contraception.
* Informed consent.

Exclusion Criteria:

* Progressed while on temozolomide.
* Evidence of acute intracranial or intratumoral hemorrhage > Grade 1.
* Not recovered from the toxic effects of prior therapy.
* Pregnant or breast feeding.
* History of diabetes mellitus.
* Uncontrolled intercurrent illness.
* Congestive heart failure, unstable angina, or a myocardial infarction within 3 months of entering the study.
* HIV positive.
* Diagnosis of another malignancy may exclude subject from study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Adverse events | 4 weeks